CLINICAL TRIAL: NCT04672512
Title: A Phase 1 Adaptive Dose, Double-Blind, Placebo-Controlled, Single and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Orally Administered CORT125329 in Healthy Subjects, With an Optional Pharmacological Effects Cohort
Brief Title: Single and Multiple Ascending Dose Study of CORT125329 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Corcept Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: CORT125329-140; 2020-001741-38 (EudraCT Number)
Record Dates: First submitted 2020-12-14; First posted 2020-12-17 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Healthy
MeSH Terms: interventions — Dosage Forms; Prednisone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- SAD Cohort A CORT125329 (Experimental): Participants will receive a single dose of CORT125329 30 mg lipid capsule formulation 1 in the fasted state on Day 1
  Interventions: Drug: CORT125329 lipid capsule formulation
- SAD Cohort B CORT125329 (Experimental): Participants will receive a single dose of CORT125329 lipid capsule formulation 1 in the fasted state on Day 1. The dose will be determined after review of safety, tolerability, and PK data from SAD Cohort A.
  Interventions: Drug: CORT125329 lipid capsule formulation
- SAD Cohorts C through H CORT125329 (Experimental): Participants will receive a single dose of CORT125329 lipid capsule formulation 1 or 2 in the fasted or fed state on Day 1 in a dose escalation format. The dose, formulation, and prandial state for each cohort will be determined after review of safety, tolerability, and PK data from previous cohorts.
  Interventions: Drug: CORT125329 lipid capsule formulation
- SAD Cohorts A through H Placebo (Placebo Comparator): Participants will receive a single dose of placebo matching CORT125329 lipid capsule formulation 1 or 2 in the fasted or fed state on Day 1 in a dose escalation format. The dose, formulation, and prandial state for each placebo cohort will match that used in the corresponding CORT125329 cohort.
  Interventions: Drug: Placebo
- MAD Cohorts A through D CORT125329 (Experimental): Participants will receive CORT125329 lipid capsule formulation 1 or 2 in the fasted or fed state on Days 1 through 14 in a dose escalation format. The dose, dose frequency (once- or twice-daily), formulation, and prandial state for each cohort will be determined after review of safety, tolerability, and PK data from previous cohorts.
  Interventions: Drug: CORT125329 lipid capsule formulation
- MAD Cohorts A through D Placebo (Placebo Comparator): Participants will receive placebo matching CORT125329 lipid capsule formulation 1 or 2 in the fasted or fed state on Days 1 through 14 in a dose escalation format. The dose, dose frequency, formulation, and prandial state for each cohort will match that used in the corresponding CORT125329 cohort.
  Interventions: Drug: Placebo
- Pharmacodynamic (PD) Effect Cohort (Experimental): Participants will receive a single dose of prednisone 25 mg in the fasted or fed state on Day 1 of Period 1. The prandial state for the Period 1 treatment will be determined after review of safety and tolerability data from the SAD Cohorts. After a 7-day washout period, participants will receive a single dose of prednisone 25 mg and a single dose of CORT125329 lipid capsule formulation 1 or 2 in the fasted or fed state on Day 1 of Period 2. The formulation and dose level of CORT125329 treatment in Period 2 will be determined after review of safety, tolerability, and PK data from the SAD cohorts. The prandial state for treatment in Period 2 will be the same used in Period 1.
  Interventions: Drug: CORT125329 lipid capsule formulation; Drug: Prednisone

INTERVENTIONS:
Drug: CORT125329 lipid capsule formulation — CORT125329 lipid capsule formulation 1 or 2 for oral administration
  Arms: MAD Cohorts A through D CORT125329; Pharmacodynamic (PD) Effect Cohort; SAD Cohort A CORT125329; SAD Cohort B CORT125329; SAD Cohorts C through H CORT125329
Drug: Placebo — Placebo matching CORT125329 lipid capsule formulation 1 or 2 for oral administration
  Arms: MAD Cohorts A through D Placebo; SAD Cohorts A through H Placebo
Drug: Prednisone — Prednisone tablet for oral administration
  Arms: Pharmacodynamic (PD) Effect Cohort

SUMMARY:
The purpose of this study is to evaluate the dose-related safety, tolerability, pharmacokinetics (PK) and pharmacological effects (PD) of CORT125329 after single and multiple ascending oral doses of CORT125329 lipid capsule formulations in healthy participants.

DETAILED DESCRIPTION:
This is a 3-part, single-center study of single and multiple ascending doses of CORT125329 in healthy participants.

Part 1 will be a double-blind, randomized, placebo-controlled assessment of single ascending doses (SAD) of CORT125329 lipid capsule formulations. Participants will be enrolled sequentially into 1 of up to 8 cohorts, each containing 8 participants.

Part 2 will be double-blind, randomized, placebo-controlled assessments of multiple oral ascending doses (MAD) of CORT125329 lipid capsule formulations. Participants will be enrolled sequentially into 1 of up to 4 cohorts, each containing 8 participants.

Optional Part 3 will be an open-label, 2-way fixed sequence cross-over study and will serve as proof of PD (glucocorticoid receptor modulation) for CORT125329 lipid capsule formulations. Participants will be enrolled in a single cohort of 10 participants.

Throughout the study, routine safety tests will be performed. In selected parts of the study, assessments of PK (CORT125329), changes in serum cortisol and plasma adrenocorticotrophic hormone (ACTH), and changes in hematological and bone biomarkers will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index of 18.0 to 30.0 kg/m^2
* Weight of ≤102 kg
* Must agree to adhere to the contraception requirements
* Additional criteria apply.

Exclusion Criteria:

* Received any investigational medicinal product in a clinical research study within the 90 days
* History of any drug or alcohol abuse in the past 2 years
* Regular alcohol consumption
* Current smokers and those who have smoked within the last 6 months
* Current users of e-cigarettes and nicotine replacement products and those who have used these products within the last 6 months
* Females of childbearing potential including those who are pregnant or lactating (all female subjects must have a negative pregnancy test at screening and admission)
* Clinically significant abnormal clinical chemistry, haematology or urinalysis as judged by the Investigator
* Confirmed positive drugs of abuse test result
* Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) results
* Active renal and/or hepatic disease
* History of clinically significant cardiovascular, renal, hepatic, endocrine, metabolic, respiratory, GI, neurological or psychiatric disorder, as judged by the Investigator
* Any form of cancer within the last 5 years (exceptions apply)
* History and/or symptoms of adrenal insufficiency
* History of clinically significant gastrointestinal disease
* Has a condition that could be aggravated by glucocorticoid antagonism
* Serious adverse reaction or serious hypersensitivity to any drug or the formulation excipients
* Presence or history of clinically significant allergy requiring treatment
* Donation or loss of greater than 400 mL of blood or plasma within the previous 3 months
* Are taking, or have taken, any prescribed, over-the-counter drug (other than 4 g per day paracetamol), vitamins or herbal remedies within 14 days before the study (exceptions may apply on a case by case basis)
* Are currently using glucocorticoids or have a history of systemic glucocorticoid use at any dose within the last 12 months or 3 months for inhaled products
* Additional criteria apply.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 115 (Actual)
Dates: Start 2020-10-23 (Actual); Primary Completion 2022-01-17 (Actual); Study Completion 2022-01-17 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with One or More Adverse Events | SAD Cohorts: up to Day 11; MAD Cohorts: up to Day 23; PD Effect Cohort: up to Day 2 in Period 1 and up to Day 11 in Period 2
Percentage of Participants with One or More Serious Adverse Events | SAD Cohorts: up to Day 11; MAD Cohorts: up to Day 23; PD Effect Cohort: up to Day 2 in Period 1 and up to Day 11 in Period 2
Percentage of Participants Discontinued from the Study Due to an Adverse Event | SAD Cohorts: up to Day 11; MAD Cohorts: up to Day 23; PD Effect Cohort: up to Day 2 in Period 1 and up to Day 11 in Period 2

SECONDARY OUTCOMES:
Plasma Pharmacokinetics (PK) of CORT125329: Maximum Observed Concentration (Cmax) | SAD Cohorts: before dosing and at prespecified time points up to Day 11; MAD Cohorts: before dosing and at prespecified time points up to Day 23; PD Effect Cohort: before dosing and at prespecified time points up to Day 11 in Period 2
Plasma PK of CORT125329: Elapsed Time from Dosing at which the Analyte was First Quantifiable in a Concentration vs Time Profile (tlag) | SAD Cohorts: before dosing and at prespecified time points up to Day 11; MAD Cohorts: before dosing and at prespecified time points up to Day 23; PD Effect Cohort: before dosing and at prespecified time points up to Day 11 in Period 2
Plasma PK of CORT125329: Time from Dosing at which Cmax was Apparent (Tmax) | SAD Cohorts: before dosing and at prespecified time points up to Day 11; MAD Cohorts: before dosing and at prespecified time points up to Day 23; PD Effect Cohort: before dosing and at prespecified time points up to Day 11 in Period 2
Plasma PK of CORT125329: Apparent Elimination Half-life (t1/2) | SAD Cohorts: before dosing and at prespecified time points up to Day 11; MAD Cohorts: before dosing and at prespecified time points up to Day 23; PD Effect Cohort: before dosing and at prespecified time points up to Day 11 in Period 2
Plasma PK of CORT125329: Area Under the Curve from Zero Time to the Last Measurable Concentration (AUC0-last) | SAD Cohorts: before dosing and at prespecified time points up to Day 11; PD Effect Cohort: before dosing and at prespecified time points up to Day 11 in Period 2
Plasma PK of CORT125329: Area Under the Curve During a Dosing Interval (AUC0-tau) | MAD Cohorts: before dosing and at prespecified time points up to Day 15
Plasma PK of CORT125329: Area Under the Curve from Zero Time Extrapolated to Infinity (AUC0-inf) | SAD Cohorts: before dosing and at prespecified time points up to Day 11; PD Effect Cohort: before dosing and at prespecified time points up to Day 11 in Period 2
Serum Cortisol | MAD Cohorts: before dosing in the morning of Days 1 and 14 and in the evening of Days -1 and 14
Plasma Adrenocorticotrophic Hormone (ACTH) | MAD Cohorts: two samples taken before dosing in the morning of Days 1 and 14 and in the evening of Days -1 and 14
Eosinophil Count | PD Effect Cohort: before dosing and at prespecified time points up to 24 hours after dosing in Period 1 and 2
Lymphocyte Count | PD Effect Cohort: before dosing and at prespecified time points up to 24 hours after dosing in Period 1 and 2
Neutrophil Count | PD Effect Cohort: before dosing and at prespecified time points up to 24 hours after dosing in Period 1 and 2
Serum Osteocalcin | PD Effect Cohort: before dosing and at prespecified time points up to 24 hours after dosing in Period 1 and 2

CONTACTS AND LOCATIONS:
Overall Officials: Sharan Sidhu, MBChB, BAO, MRCS, MFPM, Principal Investigator — Quotient Sciences
Locations (1):
- Quotient Sciences, Ruddington, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No